CLINICAL TRIAL: NCT03280654
Title: Visceral Adiposity Index and Overactive Bladder: A Novel Predictive Risk Factor
Brief Title: Visceral Adiposity Index and Overactive Bladder
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Ozan HORSANALI, Recepteutrh, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 1
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Visceral Adiposity Index
Keywords: Obesity; Overactive Bladder; Urinary incontinence; Visceral Adiposity Index; Waist Circumference
MeSH Terms: conditions — Obesity; Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:VAI levels <7,55: 7,55 value was calculated as cut-off level for VAI by ROC analyse and area under curve was calculated as 0,487 Group 1 was defined as VAI levels <7,55
  Interventions: Other: overactive bladder
- group 2:VAI levels >=7,55: 7,55 value was calculated as cut-off level for VAI by ROC analyse and area under curve was calculated as 0,487 group 2 was defined as VAI levels >=7,55
  Interventions: Other: overactive bladder

INTERVENTIONS:
Other: overactive bladder — Association between groups and over active bladder symptoms

SUMMARY:
In present study, we aimed to investigate the association between visceral adiposity index and overactive bladder symptoms in female patients aged over 18 years.Between January-2015 and July-2017, 151 female patient with overactive bladder symptoms were evaluated in Recep Tayyip Erdogan University Training and Research Hospital Urology Department. Antropometric and laboratory features including serum lipid levels, AST, ALT, fasting glucose levels, and also urodynamic findings were recorded. Visceral adiposity index was calculated according to gender-specific formula. Participants were divided into two groups according to 7,55 cut-off level for visceral adiposity index levels. Statistical significance were discussed between two groups.

DETAILED DESCRIPTION:
Antropometric and laboratory features including serum lipid levels, AST, ALT, fasting glucose levels were recorded. Urodynamic study was performed all of patients to evaluate bladder functions. Over active bladder questionnaire-8 Turkish validated short form was filled out and recorded for each patients. Detailed medical histories of all patients were obtained before the study. Height, weight, and waist circumference (WC) were measured with the subjects in their underwear. Body mass ındex (BMI) was computed by the formula as the ratio of weight to the square of height (kg/m2). WC was measured on the line between the iliac crest and the lower costal margin parallel to the ground after subjects exhaled. Inclusion criteria of study was female patients who have over active bladder symptomes with or without urinary incontinence. Exclusion criterias of study were male gender, pregnancy, alcohol intake, bladder cancer history, previous incontinence surgery history, presence of neurological disease, urinary infection or bladder stone and pelvic radiotherapy history.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 18 years aged with overactive bladder symptoms

Exclusion Criteria:

* Male gender, pregnancy, alcohol intake, bladder cancer history, previous incontinence surgery history, presence of neurological disease, urinary infection or bladder stone and pelvic radiotherapy history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with overactive bladder symptoms
Study Population: female patients over 18 years aged with overactive bladder symptoms
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Visceral adiposity index | 1 day
  Group 1(lower visceral adiposity index score) has lower over active bladder questionnaire scores than group 2(higher visceral adiposity index score)

IPD SHARING:
Plan to Share IPD: No